CLINICAL TRIAL: NCT03115476
Title: Incidence of Squamous Cell Carcinoma and Other Skin Neoplasia in Subjects With Actinic Keratosis Treated With Ingenol Disoxate Gel 0.018% or 0.037%, or Vehicle Gel
Brief Title: A Trial to Compare the Incidence of Squamous Cell Carcinoma (SCC) and Other Skin Neoplasia on Skin Areas Treated With Ingenol Disoxate Gel or Vehicle Gel for Actinic Keratosis on Face and Chest or Scalp
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined.
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LP0084-1369; 2017-000228-85 (EudraCT Number)
Record Dates: First submitted 2017-04-05; First posted 2017-04-14 (Actual); Results first posted 2019-06-25 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2019-06

CONDITIONS: Actinic Keratosis; Squamous Cell Carcinoma
MeSH Terms: conditions — Keratosis, Actinic; Carcinoma, Squamous Cell | interventions — LEO 43204

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ingenol disoxate gel 0.018% (Experimental)
  Interventions: Drug: ingenol disoxate gel 0.018%
- Ingenol disoxate gel 0.037% (Experimental)
  Interventions: Drug: ingenol disoxate gel 0.037%
- Vehicle gel (Placebo Comparator)
  Interventions: Other: Vehicle gel

INTERVENTIONS:
Drug: ingenol disoxate gel 0.018% — Ingenol disoxate gel is a novel ingenol derivative being developed for field treatment of AKs on treatment areas of up to 250 cm2 (40 in2) on the face, chest and scalp.
  Other Names: LEO 43204
  Arms: Ingenol disoxate gel 0.018%
Drug: ingenol disoxate gel 0.037% — Ingenol disoxate gel is a novel ingenol derivative being developed for field treatment of AKs on treatment areas of up to 250 cm2 (40 in2) on the face, chest and scalp.
  Other Names: LEO 43204
  Arms: Ingenol disoxate gel 0.037%
Other: Vehicle gel — Vehicle to ingenol disoxate gel with no active ingredient
  Arms: Vehicle gel

SUMMARY:
One of the main reasons for treating actinic keratoses (AK) is the wish to lower the risk of progression of AK to squamous cell carcinoma (SCC). This risk is in the order of 1 per 1000 AKs per year, which is in itself a small risk, but since patients can have dozens of AKs and the disease is chronic the cumulative risk for a patient can be substantial.

In this extension protocol of trials LP0084-1193, -1194, -1195 and -1196, LEO will study the incidence of SCCs and other skin neoplasia in vehicle and ingenol disoxate treated patients over a period of 2 years, so that the total follow-up time for each patient will be 3 years and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent has been obtained.
* The subject has been treated in one of the trials LP0084-1193, -1194, -1195, or -1196 and has been evaluated at the end of follow-up visit (month 14) of that trial.

Exclusion Criteria:

* The subject is in need of treatment with ingenol mebutate or ingenol disoxate in the selected treatment area .
* The subject is enrolled in any other interventional clinical trial.

For subjects where there is a gap between end of follow-up visit (month 14) in one of the trials LP0084-1193, -1194, -1195, or -1196 and participation in the current trial:

* The subject has been treated with ingenol mebutate or ingenol disoxate in the selected treatment area after end of follow-up visit (month 14) in one of the trials LP0084-1193, -1194, -1195, or -1196 and until participation in the current trial.
* The subject has been enrolled in any other interventional clinical trial after end of follow-up visit (month 14) in one of the trials LP0084-1193, -1194, -1195, or -1196 and until participation in the current trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (59):
- United States (30):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Dermatology Specialists, Inc, Murrieta, California
  - Dermatology Specialists, Inc., Oceanside, California
  - Contour Dermatology & Cosmetic Surgery Center, Rancho Mirage, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Therapeutics Clinical Research, San Diego, California
  - University Clinical Trials, Inc., San Diego, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - Colorado Medical Research Center, Inc., Denver, Colorado
  - AboutSkin Dermatology and DermSurgery, PC, Greenwood Village, Colorado
  - Dermatology and Dermatologic Surgery, Danbury, Connecticut
  - The GW Medical Faculty Associates, Washington D.C., District of Columbia
  - Park Avenue Dermatology, Orange Park, Florida
  - Research Institute of the Southeast, LLC, West Palm Beach, Florida
  - Visions Clincal Research, West Palm Beach, Florida
  - MedaPhase, Newnan, Georgia
  - Gwinnett Clinical Research Center, Inc., Snellville, Georgia
  - Laser & Skin Surgery Center of Indiana, Carmel, Indiana
  - Research Institute of Deaconess Clinic, Evansville, Indiana
  - DermAssociates, PC, Rockville, Maryland
  - ActivMed Practices & Research, Inc., Methuen, Massachusetts
  - Clarkston Skin Research, Clarkston, Michigan
  - Clinical Studies Group, Henderson, Nevada
  - The Dermatology Group, P.C., Verona, New Jersey
  - Skin Search of Rochester, Inc., Rochester, New York
  - Center for Clinical Studies, Houston, Texas
  - Suzanne Bruce and Associates, P.A., The Center for Skin Research, Katy, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Premier Clinical Research, Spokane, Washington
- Canada (11):
  - Investigational Site, Surrey, British Columbia
  - Investigational Site, Vancouver, British Columbia
  - Investigational Site, Winnipeg, Manitoba
  - Investigational Site, Fredericton, New Brunswick
  - Investigational Site, Ajax, Ontario
  - Investigational Site, Barrie, Ontario
  - Investigational Site, London, Ontario
  - Investigational Site, Mississauga, Ontario
  - Investigational Site, Peterborough, Ontario
  - Investigational Site, Waterloo, Ontario
  - Investigational Site, Drummondville, Quebec
- France (3):
  - Investigational Site, Chambray-lès-Tours
  - Investigational Site, Nice
  - Investigational Site, Saint-Etienne
- Germany (8):
  - Investigational Site, Berlin
  - Investigational Site, Dresden
  - Investigational Site, Frankfurt am Main
  - Investigational Site, Hamburg
  - Investigational Site, Hanover
  - Investigational Site, Münster
  - Investigational Site, Recklinghausen
  - Investigational Site, Schweinfurt
- Spain (3):
  - Investigational Site, Badalona, Barcelona
  - Investigational Site, Pamplona, Navarre
  - Investigational Site, Valencia
- United Kingdom (4):
  - Investigational Site, Dundee, Angus
  - Investigational Site, Airdrie, Lanarkshire
  - Investigational Site, Middlesbrough, North Yorkshire
  - Investigational Site, Redhill, Surrey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1234 participants were randomised and applied investigational medicinal product (IMP) in the trials LP0084-1193, -1194, -1195, -1196 (main trials, Period 1).
  A total of 563 participants from the main trials continued and were enrolled into this extension follow-up trial (LP0084-1369, Period 2).
Groups:
- Ingenol Disoxate Gel 0.018%: ingenol disoxate gel 0.018%: Ingenol disoxate gel is a novel ingenol derivative being developed for field treatment of actinic keratoses (AKs) on treatment areas of up to 250 cm2 (40 in2) on the face, chest and scalp.
- Ingenol Disoxate Gel 0.037%: ingenol disoxate gel 0.037%: Ingenol disoxate gel is a novel ingenol derivative being developed for field treatment of actinic keratoses AKs on treatment areas of up to 250 cm2 (40 in2) on the face, chest and scalp.
- Vehicle Gel: Vehicle gel to Ingenol disoxate gel with no active ingredient
Period: Main Trials (LP0084-119x)
Arm/Group | Ingenol Disoxate Gel 0.018% | Ingenol Disoxate Gel 0.037% | Vehicle Gel
Started (Total number of subjects that started in Main Trials LP0084-1193, -1194, -1195, -1196 (LP0084-119x)) | 407 | 418 | 409
Completed | 407 | 418 | 409
Not Completed | 0 | 0 | 0
Period: LP0084-1369
Arm/Group | Ingenol Disoxate Gel 0.018% | Ingenol Disoxate Gel 0.037% | Vehicle Gel
Started (Number of subjects that continued into this extension trial LP0084-1369 from the "Main trials") | 191 | 210 | 162
Completed | 0 (Trial was terminated by sponsor) | 0 (Trial was terminated by sponsor) | 0 (Trial was terminated by sponsor)
Not Completed | 191 | 210 | 162
Not completed — Death | 1 | 0 | 2
Not completed — Trial terminated by Sponsor | 190 | 210 | 160

BASELINE CHARACTERISTICS:
Population: Of the 1234 participants who were randomised and applied IMP in the Main Trials (Period1) a total of 563 participants continued into this extension follow-up trial. The endpoints in this trial are time to event endpoints, starting at randomisation in the Main Trials, and therefore the full analysis set consists of 1234 participants
Groups:
- Vehicle Gel: Vehicle gel of ingenol disoxate gel
- Total: Total of all reporting groups
Arm/Group | Ingenol Disoxate Gel 0.018% | Ingenol Disoxate Gel 0.037% | Vehicle Gel | Total
Number analyzed (Participants) | 191 | 210 | 162 | 563
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 57 | 55 | 43 | 155
  >=65 years | 134 | 155 | 119 | 408
Age, Continuous [Median (Full Range); unit: years] | 69 [48 to 88] | 71 [36 to 94] | 69 [48 to 92] | 70 [36 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 0 | 30 | 97
  Male | 124 | 210 | 132 | 466
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 3 | 0 | 12
  Not Hispanic or Latino | 182 | 206 | 162 | 550
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 190 | 209 | 162 | 561
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 43 | 62 | 53 | 158
  United States | 98 | 104 | 70 | 272
  United Kingdom | 12 | 13 | 12 | 37
  France | 2 | 6 | 4 | 12
  Germany | 19 | 25 | 17 | 61
  Spain | 17 | 0 | 6 | 23
Fitzpatrick skin type [Count of Participants; unit: Participants] — Fitzpatrick scale description:
  Type I - always burns, never tans (palest; freckles). Type II - usually burns, tans minimally Type III - sometimes mild burn, tans uniformly Type IV - burns minimally, always tans well (moderate brown) Type V - very rarely burns, tans very easily (dark brown) Type VI - never burns (deeply pigmented dark brown to darkest brown)
  Participants
    Type I | 34 | 26 | 28 | 88
    Type II | 109 | 116 | 94 | 319
    Type III | 42 | 54 | 35 | 131
    Type IV | 4 | 13 | 4 | 21
    Type V | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to First Squamous Cell Carcinoma (SCC) in the Treatment Area
Description: Time to first squamous cell carcinoma (SCC) in the treatment area. Relative difference between groups (ingenol disoxate vs vehicle) expressed as hazard ratio.
  The indicated measured values are the observed incidence rates of the SCC in the treatment area which form the basis of the statistical analysis of the time to event analysis
Time Frame: From Visit 2 (6 months after Month 14 of main trial) to first SCC in the treatment area, up to 24 months
Population: Full Analysis Set: 1234 subjects who were randomised and applied IMP in one of 4 Main Trials
Measure: Number (95% Confidence Interval); unit: SCC events per 100 patient years
Groups:
- Vehicle Gel: Vehicle gel: Ingenol disoxate gel is a novel ingenol derivative being developed for field treatment of AKs on treatment areas of up to 250 cm2 (40 in2) on the face, chest and scalp.
Arm/Group | Ingenol Disoxate Gel 0.018% | Ingenol Disoxate Gel 0.037% | Vehicle Gel
Number analyzed (Participants) | 407 | 418 | 409
SCC events per 100 patient years | 2.77 [1.55 to 4.57] | 0.88 [0.28 to 2.04] | 1.26 [0.46 to 2.74]
Statistical Analysis 1: Comparison: Ingenol Disoxate Gel 0.018% vs Ingenol Disoxate Gel 0.037% vs Vehicle Gel; Relative difference between groups (ingenol disoxate vs vehicle) expressed as hazard ratio; Test type: Other; p = 0.43, likelihood ratio test; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.61 to 3.9]

2. Secondary Outcome: Time to First Squamous Cell Carcinoma (SCC) or Other Skin Neoplasia in the Treatment Area
Description: Time to first squamous cell carcinoma (SCC) or other skin neoplasia in the treatment area. Relative difference between groups (ingenol disoxate vs vehicle) expressed as hazard ratio.
  The indicated measured values are the observed incidence rates of the SCC in the treatment area which form the basis of the statistical analysis of the time to event analysis
Time Frame: From Visit 2 (6 months after Month 14 of main trial) to first SCC or other skin neoplasia in the treatment area, up to 24 months
Population: Full Analysis Set: 1234 subjects who were randomised and applied IMP in one of 4 Main Trials
Measure: Number (95% Confidence Interval); unit: SCC events per 100 patient years
Arm/Group | Ingenol Disoxate Gel 0.018% | Ingenol Disoxate Gel 0.037% | Vehicle Gel
Number analyzed (Participants) | 407 | 418 | 409
SCC events per 100 patient years | 10.24 [7.65 to 13.4] | 2.84 [1.62 to 4.61] | 3.19 [1.79 to 5.26]
Statistical Analysis 1: Comparison: Ingenol Disoxate Gel 0.018% vs Ingenol Disoxate Gel 0.037% vs Vehicle Gel; relative difference between treatment groups (ingenol disoxate gel vs vehicle) expressed as hazard ratio; Test type: Other; p < 0.01, likelihood ratio test; Hazard Ratio (HR) = 1.99, 95% CI 2-sided [1.17 to 3.62]

ADVERSE EVENTS:
Time Frame: From first visit in this trial until the end of the trial i.e a period of up to 9 months as the trial was prematurely discontinued
Description: Only adverse events (AE) in the treatment area were collected, Serious AEs (SAE) outside treatment area were collected only if deemed related by the investigator to the study drug. This means that death not considered related to AEs in the treatment area is not included in the SAE table but are included in the All Course Mortality table For 1 subject the actual treatment was different from the planned treatment due to an error.
  Safety information is reported based on the actual treatment
Arm/Group | Ingenol Disoxate Gel 0.018% | Ingenol Disoxate Gel 0.037% | Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 1/191 | 0/211 | 2/161
Serious Adverse Events (participants affected / at risk) | 0/191 | 1/211 | 0/161
Other Adverse Events (participants affected / at risk) | 16/191 | 6/211 | 10/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ingenol Disoxate Gel 0.018% (N=191) | Ingenol Disoxate Gel 0.037% (N=211) | Vehicle Gel (N=161)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ingenol Disoxate Gel 0.018% (N=191) | Ingenol Disoxate Gel 0.037% (N=211) | Vehicle Gel (N=161)
Application site scar (General disorders) | 8 (8) | 5 (5) | 7 (7)
Application site papules (General disorders) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 1 (1)
Inflammation of wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma acknowledges the investigator right to publish the entire results of the study, irrespective of outcome. LEO Pharma retains the right to have any publication submitted to LEO Pharma for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO Pharma.

DOCUMENTS (2):
  • Study Protocol (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT03115476/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT03115476/SAP_001.pdf